CLINICAL TRIAL: NCT05048849
Title: A Phase II, Prospective, Open-Label, Multi-Center Study to Evaluate the Safety, Tolerability, and Immunogenicity of the COVID-19 Vaccine Candidate MVC-COV1901, CT-COV-21 Extension Study
Brief Title: A Study to Evaluate the Safety, Tolerability, and Immunogenicity of COVID-19 Vaccine, CT-COV-21 Extension Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medigen Vaccine Biologics Corp. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CT-COV-21e
Record Dates: First submitted 2021-09-03; First posted 2021-09-17 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2021-09

CONDITIONS: Covid19 Vaccine
Keywords: Covid19 vaccine
MeSH Terms: interventions — Adjuvants, Pharmaceutic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MVC-COV1901(S protein with adjuvant) (Experimental): S-2P protein with CpG and Aluminum Hydroxide/0.5mL
  Interventions: Biological: MVC-COV1901(S protein with adjuvant)

INTERVENTIONS:
Biological: MVC-COV1901(S protein with adjuvant) — Approximately 500 participants will receive 2 doses of MVC-COV1901(S-2P protein with adjuvant) at Day 1 and Day 29 via intramuscular (IM) injection in the deltoid region

SUMMARY:
The purpose of this study is to assess the safety and immunogenicity of MVC-COV1901 vaccine who are generally healthy or with stable pre-existing health conditions and have received 2 doses of Placebo in the main study CT-COV-21

DETAILED DESCRIPTION:
This is an extension study of the main study CT-COV-21, "A Phase II, Prospective, Double-blinded, Multi-Center, Multi-Regional Study to Evaluate the Safety, Tolerability, and Immunogenicity of the SARS-CoV-2 Vaccine Candidate MVC-COV1901."

This extension study is a prospective, open-label, multicenter study. In this extension study, approximately 500 participants who received the placebo and have remained blinded in the main study until Day 119 (90 days after the second vaccination of the main study) are enrolled and receive MVC-COV1901. Each participant will receive 2 doses of MVC-COV1901, administered 28 days apart via IM injection in the deltoid region, preferably of the non-dominant arm, at Day 1 and Day 29.

ELIGIBILITY:
Inclusion Criteria

1. Participants who are in the placebo arm of the main study (CT-COV-21), and are unblinded due to urgent condition other than safety events (i.e. on request from participants with high risk of acquiring and transmitting infection) after Day 119, are eligible.
2. Female participant must:

   1. Be either of non-childbearing potential, i.e. surgically sterilized (defined as having undergone hysterectomy and/or bilateral oophorectomy and/or bilateral salpingectomy; tubal ligation alone is not considered sufficient) or one year post-menopausal;
   2. Or, if of childbearing potential, be abstinent or agree to use medically effective contraception from 14 days before screening to 30 days following the last injection of study intervention. Acceptable forms include:

   i. Implanted hormonal methods of contraception or placement of an intrauterine device or intrauterine system ii. Established use of hormonal methods (injectable, pill, patch or ring) combined with barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository c. Have a negative pregnancy test
3. Participant is willing and able to comply with all required study visits and follow-up required by this protocol.
4. Participant or the participant's legal representative must understand the procedures of the study and provide written informed consent

Exclusion Criteria

1. Pregnant or breast feeding or have plan to become pregnant in 30 days after last administration of study intervention.
2. Employees at the investigator's site, of the Sponsor or the contract research organization (CRO) directly involved in the conduct of the study.

   Prior/Concomitant Therapy
3. Currently receiving or received any investigational intervention within 30 days prior to the first dose of study intervention.
4. Administered any licensed live-attenuated vaccines within 28 days or other licensed non-live-attenuated vaccines within 7 days prior to the first dose of study intervention.
5. Administered any blood product or intravenous immunoglobulin administration within 12 weeks prior to the first dose of study intervention.
6. Currently receiving or anticipate to receive concomitant immunosuppressive or immune-modifying therapy (excluding inhaled, topical skin and/or eye drop-containing corticosteroids, low-dose methotrexate, or < 2 weeks of daily receipt of prednisone less than 20 mg or equivalent) within 12 weeks prior to the first dose of study intervention.
7. Currently receiving or anticipate to receive treatment with tumor necrosis factor (TNF)-α inhibitors, e.g. infliximab, adalimumab, etanercept within 12 weeks prior to the first dose of study intervention.
8. Major surgery or any radiation therapy within 12 weeks prior to the first dose of study intervention
9. Participant with previous known or potential exposure to SARS-CoV-1 or 2 viruses or received any other COVID-19 vaccine.
10. Participant with a history of hypersensitivity to any vaccine or a history of allergic disease or reactions likely to be exacerbated by any component of the MVC-COV1901.
11. Body (oral, rectal, or ear) temperature ≥ 38.0°C or acute illness (not including minor illnesses such as diarrhea or mild upper respiratory tract infection at the discretion of the investigator) within 2 days before the first dose of study intervention.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2021-07-19 (Actual); Primary Completion 2021-11-08 (Actual); Study Completion 2022-04-12 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Event (Safety of MVC-COV1901) | Day 1 to 28 days after second vaccination
  To evaluate the safety and tolerability of MVC-COV1901 from Day 1 to 28 days after the second dose of study intervention in terms of the number of participants with the occurrence of:
  * Solicited local AEs (up to 7 days after each dose of study intervention)
  * Solicited systemic AEs (up to 7 days after each dose of study intervention)
  * Unsolicited AEs (up to 28 days after each dose of study intervention)
  * AE of Special Interest (AESI)
  * Vaccine-Associated Enhanced Disease(VAED)
  * Serious adverse events (SAEs)
Percentage of Adverse Event (Safety of MVC-COV1901) | Day 1 to 28 days after second vaccination
  To evaluate the safety and tolerability of MVC-COV1901 from Day 1 to 28 days after the second dose of study intervention in terms of the percentage of participants with the occurrence of:
  * Solicited local AEs (up to 7 days after each dose of study intervention)
  * Solicited systemic AEs (up to 7 days after each dose of study intervention)
  * Unsolicited AEs (up to 28 days after each dose of study intervention)
  * AE of Special Interest (AESI)
  * Vaccine-Associated Enhanced Disease(VAED)
  * Serious adverse events (SAEs)
Immunogenicity of MVC-COV1901(Neutralizing Antibody) | Day 1 to 28 days after second vaccination
  To evaluate the immunogenicity of MVC-COV1901 in terms of neutralizing antibody titers 28 days after the second dose of study intervention

SECONDARY OUTCOMES:
Number of Adverse Event over the study period (Secondary Safety of MVC-COV1901) | Day 1 to 180 days after second vaccination
  To evaluate the safety of MVC-COV1901 over the study period in terms of the number of participants with the occurrence of:
  * >= Grade 3 AE
  * AE of Special Interest (AESI)
  * Vaccine-Associated Enhanced Disease(VAED)
  * Serious adverse events (SAEs)
Percentage of Adverse Event over the study period (Secondary Safety of MVC-COV1901) | Day 1 to 180 days after second vaccination
  To evaluate the safety of MVC-COV1901 over the study period in terms of the percentage of participants with the occurrence of:
  * >= Grade 3 AE
  * AE of Special Interest (AESI)
  * Vaccine-Associated Enhanced Disease(VAED)
  * Serious adverse events (SAEs)
Immunogenicity of MVC-COV1901(Antigen-specific Immunoglobulin) | Day 1 to 28 days after second vaccination
  To evaluate the immunogenicity of MVC-COV1901 in terms of antigen-specific immunoglobulin 28 days after the second dose of study intervention

OTHER OUTCOMES:
Incidence of confirmed COVID-19 cases (Efficacy of MVC-COV1901) | Day 1 to 180 days after second vaccination
  To estimate the efficacy of MVC-COV1901, as compared to placebo, in the prevention of COVID-19 in terms of :
  * The number of laboratory-confirmed COVID-19 cases occurring ≥ 15 days after any dose of study intervention.
  * The number of laboratory-confirmed COVID-19 severe cases occurring ≥ 15 days after any dose of study intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Szu-Min Hsieh, MD, Principal Investigator — National Taiwan University Hospital; Tzou-Yien Lin, MD, Principal Investigator — Chang Gang Memorial Hospital, LinKou
Locations (11):
- Taiwan (11):
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Taipei Municipal Wan Fang Hospital, Taipei
  - Taipei Veteran General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang-Guang Memorial Hospital Lin-Kou, Taoyuan District
  - Tao-Yuan General Hospital, Taoyuan District

IPD SHARING:
Plan to Share IPD: No